CLINICAL TRIAL: NCT02402205
Title: TF-CBT for Adjudicated Youth in Residential Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Judith Cohen, Medical Director, Professor of Psychiatry, Allegheny General Hospital, Drexel University College of Medicine, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: R01MH095208 (NIH)
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: PTSD
Keywords: Implementation; TF-CBT; adjudicated youth; RTF; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web Implementation of TF-CBT (Experimental): Web implementation ("W")provides only web-based (distance learning) training and consultation to mental health therapists providing TF-CBT treatment to adjudicated youth in RTF. Therapists access the initial 10 hour training course(www.musc.edu/tfcbt) and follow-up consultation (www.musc.edu/tfcbtconsult) at their own convenience and as needed during the course of the study, with RTF administrators guaranteeing that therapists have time to do so. This implementation strategy is free and more convenient to therapists and administrators as it can be accessed whenever desired.
  Interventions: Behavioral: TF-CBT
- Web + Live Implementation of TF-CBT (Experimental): Web + Live ("W+L") implementation provides web-based training and consultation as described in W, and also provides 1) face-to-face training and 2) twice monthly phone consultation with an expert TF-CBT trainer. W+L requires greater resource commitment from therapists and administrators and is less convenient, but provides more specific consultation on the therapists' personal TF-CBT treatment cases.
  Interventions: Behavioral: TF-CBT

INTERVENTIONS:
Behavioral: TF-CBT — Web TF-CBT implementation or Web + Live TF-CBT implementation

SUMMARY:
Adjudicated youth often have traumatic stress responses but rarely receive treatment for these problems. This study is a randomized controlled trial to evaluate two alternative implementation strategies for providing an evidence-based trauma treatment, Trauma-Focused Cognitive Behavioral Therapy (TF-CBT), to therapist who treat adjudicated youth in 18 residential treatment facilities (RTF) in New Hampshire, Vermont, and Connecticut: 1) web-based TF-CBT implementation strategy ("W"), consisting on only web-based training and consultation; versus 2) W plus live TF-CBT implementation strategy, consisting of W plus face-to face training and phone consultation with TF-CBT experts ("W+L").

DETAILED DESCRIPTION:
Therapists in each of 18 participating RTFprograms that serve adjudicated youth are randomized to receive either:

1. W TF-CBT implementation strategy, provided via the free distance learning resources TF-CBTWeb, (www.musc/edu/tfcbt) and TF-CBTConsult (www.musc.edu/tfcbtconsult); or
2. W+L implementation strategy, provided through W + 2 day TF-CBT training plus one year of twice monthly TF-CBT consultation calls with a TF-CBT expert trainer.

All RTF staff receive one day training in trauma-informed care. All therapists in both conditions receive training in screening youth for trauma exposure and symptoms. Data are collected regarding primary outcomes of: 1) number of youth therapists in each condition screen for trauma symptoms, 2) number of youth consent to TF-CBT treatment; 3) number of youth complete TF-CBT, 4) TF-CBT fidelity during treatment. Secondary outcomes include 1)changes in therapist knowledge and satisfaction regarding TF-CBT treatment and 2) youth outcomes including PTSD symptoms, depression and satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria: Consenting mental health therapists in participating residential treatment facilities (RTF)in New Hampshire, Vermont and Connecticut; and the adjudicated youth ages 12-17 years old who are residents in these RTF programs being treated by the participating therapists who 1) are screened positive for having at least one past trauma experience with UCLA PTSD Reaction Index score of >22; 2) assent with legal guardian consent to participate in the project; and 3) are anticipated to remain in the RTF program at least 3 months (long enough to receive TF-CBT treatment).

-

Exclusion Criteria: Guardian or youth refuses;youth does not endorse trauma exposure or symptoms; youth is being discharged too soon to participate; Therapist may use clinical judgment to exclude youth from study based on clinical presentation.

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of youth screened for trauma exposure and PTSD symptoms | Day 1
  Number of youth screened for trauma exposure and PTSD symptoms using the UCLA PTSD Reaction Index (online version)in W vs. W+L implementation condition
Number of youth starting TF-CBT | Day 60
  Number of youth who begin TF-CBT treatment in W vs W+L implementation condition
Number of youth completing TF-CBT in each condition | Day 240 (6 months post start of treatment)
  Number of youth completing TF-CBT in W vs W+L conditions
Fidelity of TF-CBT implementation | Day 240
  Therapist fidelity implementing TF-CBT across and between implementation conditions using TF-CBT Fidelity Checklist (online version)

SECONDARY OUTCOMES:
Therapy Procedures Checklist | Day 1; Day 900 (30 monhts later)
  Therapist comfort with cognitive therapy practices (or change in this during the study) as a predictor of other outcomes between the W vs. W+L group
Attitudes toward Computer Usage Scale | Day 1; Day 900
  Attitudes toward computer usage as a potential covariate of outcomes
TF-CBTWeb Knowledge Test | Day 1, Day 900
  Change in knowledge related to TF-CBT as a moderator of outcomes
Youth UCLA PTSD Reaction Index | Day 1; Day 240 (post treatment_
  Change in youth PTSD scores across and between implementation conditions to be examined as a secondary outcome
Mood and Feelings Questionnaire-Short Version | Day 1; Day 240 (post treatment)
  Change in youth depression scores in youth across and between implementation conditions
Youth Satisfaction Survey | Day 240 (post treatment)
  Youth satisfaction with therapy across and between implementation conditions

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Cohen, M.D., Principal Investigator — West Penn Allegheny Health System